CLINICAL TRIAL: NCT06534411
Title: Efficacy and Safety of Co-administered Cagrilintide and Semaglutide (CagriSema) 1.0 mg/1.0 mg s.c. Once Weekly Versus Tirzepatide 5 mg s.c. Once Weekly in Participants With Type 2 Diabetes Inadequately Controlled on Metformin, SGLT2 Inhibitor or Both
Brief Title: A Research Study to See How Much CagriSema Lowers Blood Sugar and Body Weight Compared to Tirzepatide in People With Type 2 Diabetes Treated With Metformin, SGLT2 Inhibitor or Both
Acronym: REIMAGINE 5
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9388-7741; U1111-1300-2590 (Other: World Health Organization (WHO)); 2023-509600-15 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — cagrilintide; semaglutide; Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CagriSema (Experimental): Participants will receive once-weekly subcutaneous (s.c) injections of CagriSema (cagrilintide and semaglutide) at escalating doses every 4 weeks in a 8-week dose escalation period until target dose of CagriSema is achieved and maintained for 52 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Tirzepatide (Experimental): Participants will receive once-weekly s.c injections of tirzepatide at escalating dose in a 4-week dose escalating period and maintained up to 56 weeks.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Cagrilintide — Participants will receive once-weekly cagrilintide subcutaneously.
  Arms: CagriSema
Drug: Semaglutide — Participants will receive once-weekly semaglutide subcutaneously.
  Arms: CagriSema
Drug: Tirzepatide — Participants will receive once-weekly tirzepatide subcutaneously.
  Arms: Tirzepatide

SUMMARY:
This study will look at how much CagriSema lowers blood sugar and body weight in people with type 2 diabetes. CagriSema is a new investigational medicine. Doctors cannot yet prescribe CagriSema. CagriSema will be compared to a medicine called tirzepatide. Doctors can prescribe tirzepatide in some countries. Participants will either receive CagriSema or tirzepatide. Which treatment the participant will receive is decided by chance. For each participant, the study will last for up to 1 year and 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (sex at birth).
* Age 18 years or above at the time of signing the informed consent.
* Diagnosed with type 2 diabetes mellitus greater than or equal to (>=) 180 days before screening.
* Stable daily dose(s) >= 90 days before screening of any of the following antidiabetic drug(s) or combination regimen(s) at effective or maximum tolerated dose as judged by the investigator:
* Metformin
* sodium-glucose co-transporter 2 inhibitor (SGLT2i)
* Glycated haemoglobin (HbA1c) 7.0-10.5 percent (53-91 millimoles per mol [mmol/mol]) (both inclusive) as determined by central laboratory at screening.
* Body mass index (BMI) >= 30 kilogram per square meter (kg/m^2) at screening. BMI will be calculated in the electronic case report form (eCRF) based on height and body weight at screening.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using a highly effective contraceptive method.
* Renal impairment with estimated Glomerular Filtration Rate less than < 30 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) as determined by central laboratory at screening.
* Treatment with any anti-diabetic or anti-obesity medication (irrespective of indication) other than stated in the inclusion criteria within 90 days before screening. However, short term insulin treatment for a maximum of 14 consecutive days is allowed.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by an eye examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1023 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-07-14 (Estimated)

PRIMARY OUTCOMES:
Change in Glycated Haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 60)
  Measured in percentage points.
Relative Change in Body Weight | From baseline (week 0) to end of treatment (week 60)
  Measured in percentage (%).

SECONDARY OUTCOMES:
Change in HbA1c | From baseline (week 0) to end of treatment (week 60)
  Measured in percentage points.
Change in Fasting Plasma Glucose (FPG) | From baseline (week 0) to end of treatment (week 60)
  Measured as millimole per liter (mmol/L).
Number of Participants Who Achieve HbA1c Target Values of Less Than (<) 7.0 (Percent [%]) (< 53 millimole per mole [mmol/mol]) | At end of treatment (week 60)
  Measured as count of participants.
Number of Participants Who Achieve HbA1c Target Values of Less Than or Equal to (<=) 6.5% (<= 48 mmol/mol) | At end of treatment (week 60)
  Measured as count of participants.
Number of Participants Who Achieve Greater Than or Equal to (>=) 5% Weight Reduction | From baseline (week 0) to end of treatment (week 60)
  Measured as count of participants.
Number of Participants Who Achieve >= 10% Weight Reduction | From baseline (week 0) to end of treatment (week 60)
  Measured as count of participants.
Number of Participants Who Achieve >= 15% Weight Reduction | From baseline (week 0) to end of treatment (week 60)
  Measured as count of participants.
Number of Participants Who Achieve >= 20% Weight Reduction | From baseline (week 0) to end of treatment (week 60)
  Measured as count of participants.
Change in Systolic Blood Pressure (SBP) | From baseline (week 0) to end of treatment (week 60)
  Measured in millimeter of mercury (mmHg).
Change in Diastolic Blood Pressure (DBP) | From baseline (week 0) to end of treatment (week 60)
  Measured in mmHg.
Change in Waist Circumference | From baseline (week 0) to end of treatment (week 60)
  Measured in centimeter (cm).
Ratio to Baseline in Lipids: Total Cholesterol | From baseline (week 0) to end of treatment (week 60)
  Measured as ratio.
Ratio to Baseline in Lipids: High Density Lipoprotein (HDL) Cholesterol | From baseline (week 0) to end of treatment (week 60)
  Measured as ratio.
Ratio to Baseline in Lipids: Low Density Lipoprotein (LDL) Cholesterol | From baseline (week 0) to end of treatment (week 60)
  Measured as ratio.
Ratio to Baseline in Lipids: Very Low Density Lipoprotein (VLDL) Cholesterol | From baseline (week 0) to end of treatment (week 60)
  Measured as ratio.
Ratio to Baseline in Lipids: Triglycerides | From baseline (week 0) to end of treatment (week 60)
  Measured as ratio.
Ratio to Baseline in Lipids: Non-HDL cholesterol | From baseline (week 0) to end of treatment (week 60)
  Measured as ratio.
Change in Short Form (SF) -36v2 Score: Physical Component Summary Score | From baseline (week 0) to end of treatment (week 60)
  Measured as score points. SF-36v2 Acute measures Health-Related Quality of Life (HRQOL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2. Acute scores are norm-based scores, i.e. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Physical component summary scores ranges from 6.1 to 79.7 with higher scores indicating better functional health and well-being.
Change in SF-36v2 Score: Mental Component Summary Score | From baseline (week 0) to end of treatment (week 60)
  Measured as score points. SF-36v2 Acute measures Health-Related Quality of Life (HRQOL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2. Acute scores are norm-based scores, i.e. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Mental component summary scores ranges from -3.8 to 78.7 with higher scores indicating better functional health and well-being.
Change in SF-36v2 Score: Vitality Subscale | From baseline (week 0) to end of treatment (week 60)
  Measured as score points. SF-36v2 Acute measures Health-Related Quality of Life (HRQOL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2. Acute scores are norm-based scores, i.e. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Vitality score ranges from 25.6 to 69.1 with higher scores indicating better functional health and well-being.
Change in Impact of Weight on Quality of Life Lite for Clinical Trials Version (IWQOL-Lite-CT) : Physical Function score | From baseline (week 0) to end of treatment (week 60)
  Measured as score points. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. Physical functioning score ranges from 0 to 100, with higher scores reflecting better levels of functioning.
Change in IWQOL-Lite-CT: Total score | From baseline (week 0) to end of treatment (week 60)
  Measured as score points. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. Total score ranges from 0 to 100, with higher scores reflecting better levels of functioning.
Number of Treatment Emergent Adverse Events (TEAEs) | From baseline (week 0) to end of study (week 66)
  Measured as count of events.
Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (<54 Milligram per Deciliter [mg/dL]), Confirmed by Blood Glucose (BG) Meter | From baseline (week 0) to end of study (week 66)
  Measured as count of episodes.
Number of Severe Hypoglycaemic Episodes (Level 3): Hypoglycaemia Associated With Severe Cognitive Impairment Requiring External Assistance for Recovery, With no Specific Glucose Threshold | From baseline (week 0) to end of study (week 66)
  Measured as count of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (162):
- United States (54):
  - Cahaba Research, Pelham, Alabama
  - Velocity Clinical Research-Phoenix, Phoenix, Arizona
  - AES Tucson DRS, Tucson, Arizona
  - Woodland Int. Research Group, Little Rock, Arkansas
  - Velocity Clin Res-Chula Vista, Chula Vista, California
  - John Muir Physicians Network, Concord, California
  - Diabetes & Endocrine Specialists - La Mesa, La Mesa, California
  - Velocity Clin Research LA, Los Angeles, California
  - Desert Oasis Healthcare, Palm Springs, California
  - Velocity Clin Res Santa Ana, Santa Ana, California
  - Velocity Clin Res - Panorama, Van Nuys, California
  - Optumcare Clinical Trials,LLC-Golden, Colorado Springs, Colorado
  - FEME Medical LLC, Washington D.C., District of Columbia
  - Tampa Bay Medical Research, Clearwater, Florida
  - AGA Clinical Trial, Hialeah, Florida
  - Clinical Trial Services Corp, Miami, Florida
  - Bioclinical Research Alliance, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - South Broward Research LLC, Miramar, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Optimal Research Sites, Orange City, Florida
  - Javara Inc. / Privia Medical Group Georgia LLC, Fayetteville, Georgia
  - Clinical Invest Special_Gurnee, Gurnee, Illinois
  - Iowa Diabetes & Endo Res Ctr, West Des Moines, Iowa
  - Cotton-Oneill Diabetes and End, Topeka, Kansas
  - AES Minneapolis DRS, Richfield, Minnesota
  - Velocity Clin Res Gulfport, Gulfport, Mississippi
  - AES St. Louis DRS, St Louis, Missouri
  - Univ of Nebraska Medical CTR, Omaha, Nebraska
  - Velocity Clin Res Albuquerque, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Carteret Medical Group, Morehead City, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Triad Research Institute, Norman, Oklahoma
  - Circuit Clinical - PMSI, Pottstown, Pennsylvania
  - Clinical Res Collaborative, Cumberland, Rhode Island
  - Velocity Clin Res Providence, East Greenwich, Rhode Island
  - Velocity Clin Res Gaffney, Gaffney, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Clinical Research Associates, Nashville, Tennessee
  - Velocity Clin Res Austin, Austin, Texas
  - AES Dallas DFW DRS, Dallas, Texas
  - UT Southwestern Medical Center - Lingvay, Dallas, Texas
  - JCCT- Juno NW Houston, Houston, Texas
  - Discovery MM Services - Houston - Broadway Street, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Aeres Clinical Research, Laredo, Texas
  - RGV Endocrine Center, McAllen, Texas
  - Privia Health Javara Clin Res., Stephenville, Texas
  - J.Lewis Research Inc, Salt Lake City, Utah
  - Chrysalis Clinical Research, St. George, Utah
  - TPMG Clinical Research, Newport News, Virginia
- Argentina (7):
  - Centro Médico CIMEL, Lanús Este, Buenos Aires
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata, Buenos Aires
  - Fundación CESIM, Santa Rosa, La Pampa Province
  - Centro de Investigaciones Médicas Tucumán, San Miguel de Tucuimán, Tucumán Province
  - IMOBA, City of Buenos Aires
  - Centro de Investigaciones Metabólicas, City of Buenos Aires
  - Instituto de Investigaciones Clinicas San Nicolás, San Nicolás
- Australia (7):
  - Paratus Clinical, Bruce, Australian Capital Territory
  - Hunter Diabetes Centre, Merewether, New South Wales
  - Austrials, St Leonards, New South Wales
  - Momentum Clinical Research, St Leonards, New South Wales
  - Roger Chih Yu Chen, Sydney, New South Wales
  - Townsville University Hospital, Douglas, Queensland
  - Paratus Clinical, Herston, Queensland
- Brazil (3):
  - Centro de Diabetes Curitiba, Curitiba, Paraná
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul Ltda., Porto Alegre, Rio Grande do Sul
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
- Canada (13):
  - Hilltop Medical Clinic, Surrey, British Columbia
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Centricity Research Brampton, Brampton, Ontario
  - Centricity Research Etobicoke, Etobicoke, Ontario
  - Wharton Med Clin Trials, Hamilton, Ontario
  - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Ctr de rech Clin de Laval, Laval, Quebec
  - Alpha Recherche Clinique - Clinique de Levis, Lévis, Quebec
  - Centre Medical Acadie, Montreal, Quebec
  - Ctr de Med Metab de Lanaudiere, Terrebonne, Quebec
  - Diex Recherche Victoriaville, Victoriaville, Quebec
  - Centre de Recherche Saint-Louis, Québec
- Germany (8):
  - Herz- und Diabeteszentrum NRW - Bad Oeynhausen, Bad Oeynhausen
  - Universitätsklinikum Essen - Klinik für Endokrinologie, Diabetologie und Stoffwechsel, Essen
  - Praxis am Markt Dr. Becker, Essen
  - Universitätsklinikum Freiburg - Innere Medizin II, Freiburg im Breisgau
  - Wendisch/Dahl Hamburg (DZHW), Hamburg
  - Medicover Neuroendokrinologie MVZ München, München
  - MedicalCenter am Clemenshospital - Schwerpunktpraxis für Diabetologie und Ernährungsmedizin, Münster
  - Zentrum für klinische Studien Allgäu Oberschwaben, Wangen
- Greece (8):
  - Alexandra General Hospital, Therapeutic Clinic, Athens, Attica
  - General Hospital Venizeleio-Pananeio - Diabetic Clinic, Heraklion, Crete
  - Evangelismos Hospital, Athens
  - Iatriko Athinon 'Palaiou Falirou', Athens
  - "Laiko" General Hospital of Athens, Goudi/Athens
  - University General Hospital of Ioannina,Internal Medicine, Ioannina
  - General Hospital of Thessaloniki 'G. Gennimatas, Thessaloniki
  - 'Ippokrateio' General Hospital of Thessaloniki, Thessaloniki
- Hungary (10):
  - Szegedi Tudomanyegyetem St Györgyi Albert Klinikai Központ, Szeged, Csongrád-Csanád
  - Komáromi Selye János Kórház, Komárom, Komárom-Esztergom
  - QUALICLINIC Egészségügyi Szolgáltató és Kutatásszervező Kft, Budapest, Pest County
  - Óbudai Egészségügyi Centrum, Budapest, Pest County
  - Szőcs Depot Egészségügyi Szolgáltató Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - ClinDiab Egészségügyi Szolgáltató és Kereskedelmi Kft., Budapest
  - PVN Kutato Kft., Budapest
  - MED-TIMA Kft., Budapest
  - Észak-Pesti Centrumkórház Honvédkórház, Budapest
- India (13):
  - Endolife Specialty Hospitals, Guntur, Andhra Pradesh
  - Ramaiah Memorial Hospital, Bengaluru, Karnataka
  - Excel Endocrine Centre, Kolhāpur, Maharashtra
  - Acharya Vinoba Bhave Rural Hospital, Sawangi Meghe, Wardha, Wardha, Maharashtra
  - All India Institute of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi
  - Jawahar Lal Nehru Govt. Medical College, Ajmer, Rajasthan
  - SMS Hospital, Jaipur, Rajasthan
  - Diabetes, Thyroid and Endocrine Centre, Jaipur, Rajasthan
  - Arthur Asirvatham hospital,, Madurai, Tamil Nadu
  - Jawaharlal Institute of Postgraduate Medical Education and Research (JIPMER), Puducherry, Tamil Nadu
  - AIG Hospitals,Hyderabad, Hyderabad, Telangana
  - Udyaan Health Care, Lucknow, Uttar Pradesh
  - IPGME&R and SSKM Hospital, Kolkata, West Bengal
- Israel (7):
  - Clalit sick fund Herzeliya, Herzeliya, Israel
  - Rambam MC - Diabetes and obesity center of excellence, Haifa
  - Wolfson MC - Diabetes Clinic, Holon
  - Hadassah Ein Karam MC - Diabetes Unit, Jerusalem
  - Rabin MC Beilinson - Endo unit, Petah Tikva
  - Sourasky MC - Institute of Endocrinology, metabolism and hypertension, Tel Aviv
  - Sheba MC - Endocrinology Clinic, Tel Litwinsky
- Poland (9):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Diab Serwis Popenda Spółka Jawna, Chorzów
  - Specjalistyczny Gabinet Diabetologiczny Rumianowski Radosław, Gorzów Wielkopolski
  - Centrum Terapii Wspolczesnej - J.M. Jasnorzewska S.K.A., Lodz
  - Etyka Osrodek Badan Klinicznych Tomasz Pesta S.K.A., Olsztyn
  - Kiepury Clinic MALGORZATA JARNOT SPECJALISTYCZNA PRAKTYKA GINEKOLOGICZNO-POLOZNICZA, Sosnowiec
  - Centrum Medyczne Oporow, Wroclaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. Prof. Szyszko, Zabrze
- Romania (8):
  - Diabdana S.R.L., Oradea, Bihor County
  - Institutul National De Diabet Nutritie Si Boli Metabolice Prof.Dr.N.Paulescu Bucuresti- Ion Movila, Bucharest, Bucurestii
  - CMI Dr Pop Lavinia, Baia Mare, Maramureş
  - Sc Mediab Srl, Târgu Mureş, Mureș County
  - SC Nutrilife SRL, Bucharest
  - Diabet Med SRL, Bucharest
  - Sanamed Hospital SRL, Bucharest
  - Clinica Korall S.R.L. Satu Mare, Satu Mare
- Spain (6):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Centro Periferico De Especialidades Bola Azul, Almería
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario San Cecilio, Granada
  - Clínica Nuevas Tecnologías en Diabetes y Endocrinología, Seville
  - Hospital Clínico de Valladolid, Valladolid
- Taiwan (9):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaoshiung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou, Taoyuan
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisktrials.com
URL: https://novonordisk-trials.com